CLINICAL STUDY PROTOCOL
PROTOCOL NUMBER: 43USD1802

#### CONFIDENTIAL

#### This document contains confidential, proprietary information

All the information provided to the Investigator and his/her staff and all data obtained through this Q-Med AB clinical study protocol are confidential. The Sponsor reserves all proprietary rights. No information may be disclosed to any third party without prior written consent from Q-Med AB.



#### **TITLE PAGE**

Dysport Efficacy and Measured Satisfaction (DREAM) Study: A Multicenter, Open-Label, Interventional Study to Evaluate Subject Satisfaction of AbobotulinumtoxinA Treatments in Moderate to Severe Glabellar Lines

> CTN: 43USD1802 Protocol Amendment 1

#### **SPONSOR:**

Name: Q-Med AB, a Nestlé Skin Health affiliate

Address:

Phone:

#### **CONTRACT RESEARCH ORGANIZATION (CRO):**

Name: MedTrials, Inc.

Address:

Phone:

#### **SAFETY:**

For safety questions, please contact the Sponsor Contact using the contact details provided in Section 12.9. Serious adverse events (SAEs) and pregnancy report forms should be submitted as described in Sections 8.2.1.2.2 and 8.2.1.2.3.

#### **MEDICAL MONITOR:**

For any medical questions related to the clinical study protocol, please contact the Medical Monitor using the contact details provided in Section 12.9.

This clinical study shall be performed in compliance with the clinical trial agreement (CTA), the CSP, ICH-Good Clinical Practice (GCP), and applicable regional and national regulations. The study shall be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki (https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/).



## **Table of Contents**

| ~~~~ | LE PAGE | |
|---|---|---|
| SYN | OPSIS | 8 |
| CLI | NICAL STUDY SCHEMATIC AND FLOW CHART | 13 |
| SCH | IEDULE OF ASSESSMENTS | 15 |
| LIST | Γ OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 17 |
| 1 | BACKGROUND AND RATIONALE | 19 |
| 1.1 | Medical Background and Short Rationale for the Clinical Study | 19 |
| 1.2 | Drug Profile | 19 |
| 1.3 | Risk/Benefit Assessment | 20 |
| 2 | CLINICAL STUDY OBJECTIVES AND CLINICAL HYPOTHESIS | 20 |
| 2.1 | Clinical Study Objectives | 20 |
| 2.1.1 | Primary Efficacy Objectives and Endpoints | 21 |
| 2.1.3 | Safety Objectives and Endpoints | 22 |
| 3 | | |
| 5.1 | Number of Subjects | 23 |
| 5.1<br>5.2 | Number of Subjects Clinical Study Population Characteristics | |
| | Clinical Study Population Characteristics | 23 |
| 5.2 | Clinical Study Population Characteristics Inclusion Criteria | 23 |
| 5.2<br>5.2.1 | Clinical Study Population Characteristics Inclusion Criteria | 23<br>23 |
| <ul><li>5.2</li><li>5.2.1</li><li>5.2.2</li></ul> | Clinical Study Population Characteristics Inclusion Criteria Exclusion Criteria | 232324 |
| <ul><li>5.2</li><li>5.2.1</li><li>5.2.2</li><li>5.3</li></ul> | Clinical Study Population Characteristics | 232324 |
| <ul><li>5.2</li><li>5.2.1</li><li>5.2.2</li><li>5.3</li></ul> | Clinical Study Population Characteristics | 23<br>23<br>24 |
| <ul><li>5.2</li><li>5.2.1</li><li>5.2.2</li><li>5.3</li></ul> | Clinical Study Population Characteristics | 232324 |
| <ul><li>5.2</li><li>5.2.1</li><li>5.2.2</li><li>5.3</li></ul> | Clinical Study Population Characteristics | 23<br>23<br>24 |

| 5.5 | Procedures/Reasons for Subject Discontinuation | 27 |
|-------|----------------------------------------------------|----|
| 6 | CLINICAL SUPPLIES | 29 |
| 6.1 | Clinical Supply Identification and Use | 29 |
| 6.1.2 | Subject Identification Number (SIN) | 29 |
| 6.1.3 | Method of Treatment Assignment | 30 |
| 6.1.4 | Kit Number/Randomization Number | 30 |
| 6.3.3 | B Dispensing and Return | 33 |
| 6.3.4 | Treatment Compliance Management and Record | 33 |
| 6.4 | Dose Modification | 33 |
| 6.5 | Blinding | 33 |
| 7 | EFFICACY ASSESSMENTS | 34 |
| 7.1 | Overall Subject Satisfaction by Direct Questioning | 34 |
| 8 | SAFETY ASSESSMENTS | 36 |
| 8.1 | Focused Physical Examination | 36 |
| 8 2 | Adverse Events | 36 |

| 8.2.1.1 | <b>Definitions</b> | 36 |
|---|---|---|
| 8.2.1.1.1 | Adverse Events (AE) | 36 |
| 8.2.1.1.2 | Treatment Emergent Adverse Events (TEAE) | 37 |
| 8.2.1.1.3 | Serious Adverse Events (SAE) | 37 |
| 8.2.1.1.4 | Unexpected Adverse Drug Reaction | 38 |
| 8.2.1.1.5 | Adverse Event Reporting Period | 38 |
| 8.2.1.1.6 | Severity | 38 |
| 8.2.1.1.7 | Relationship to the Study Product and/or Clinical Study Procedure | 38 |
| 8.2.1.2 | Reporting Procedures | 39 |
| 8.2.1.2.1 | Procedures for Reporting Adverse Events | 39 |
| 8.2.1.2.2 | Procedure for Reporting a Serious Adverse Event | 40 |
| 8.2.1.2.3 | Procedures for Reporting Pregnancies | 41 |
| 8.3 O | Other Assessments | 42 |
| 8.3.2 | Pregnancy Test | 42 |
| 8.4 A | Appropriateness of Measurements | 42 |
| 9 CLI | NICAL STUDY VISITS DESCRIPTIONS AND PROCEDURES | 43 |
| | | 48 |
| 10 STA | TISTICAL METHODS PLANNED | 49 |

| 10.1.2.4 | Safety Population | 49 |
|----------|------------------------------------------------------------|----|
| 10.1.2.5 | Imputation of Missing Data | 50 |
| 10.1.3.1 | Safety | 50 |
| 10.1.4 | Withdrawals and Deviations | 51 |
| 10.1.5 | | |
| 11 T | RAINING / MONITORING / DATA MANAGEMENT / QUALITY ASSURANCE | 52 |
| 11.1 | Personnel Training | 52 |
| 11.2 | Clinical Monitoring | 52 |
| 11.3 | Data Management | 52 |
| 11.4 | Quality Assurance / Audit / Inspection | 52 |
| 12 E | THICS AND GENERAL CLINICAL TRIAL CONDUCT CONSIDERATIONS | 54 |
| 12.1 | Institutional Review Board (IRB) | 54 |
| 12.2 | Ethical Conduct of the Clinical Study | 54 |
| 12.3 | Subject Information and Consent | 54 |
| 12.4 | Protection of Personal Data | 54 |
| 12.5 | Contractual Requirements | 55 |
| 12.6 | Data Collection and Archiving | 55 |
| 12.6.1 | Data Collection | 55 |
| 12.6.2 | Source Documentation | 55 |
| 12.6.3 | Archives | 56 |
| 12.7 | Insurance | 56 |





| 13 | LITERATURE REFERENCE LIST | <b>58</b> |
|----|---------------------------|------------|
| 14 | APPENDICES | <b>5</b> 9 |
| | | _ |
| | List of Tables | |
| | List of Figures | |





# **SYNOPSIS** Clinical Study Title: Dysport Efficacy and Measured Satisfaction (DREAM) Study: A Multicenter, Open-Label, Interventional Study to Evaluate Subject Satisfaction of AbobotulinumtoxinA Treatments in Moderate to Severe Glabellar Lines or Female of childbearing potential with a negative urine pregnancy test at screening/baseline, and agrees to use an acceptable, reliable and approved contraceptive method for the duration of enrollment in the study. Male subjects do not require birth control measures. Time and ability to complete the study and comply with instructions. 6. Understands the study requirements and signed the informed consent form (ICF). **Key Exclusion Criteria** Botulinum toxin treatment in the face within 9 months prior to the screening/baseline visit. Known allergy or sensitivity to any component of the study product, or allergy to cow's milk protein.







## **SYNOPSIS** Clinical Study Title: Dysport Efficacy and Measured Satisfaction (DREAM) Study: A Multicenter, Open-Label, Interventional Study to Evaluate Subject Satisfaction of AbobotulinumtoxinA Treatments in Moderate to Severe Glabellar Lines The primary endpoint will evaluate the proportion of subjects satisfied ("highly satisfied" or "satisfied") with the treatment results assessed by the satisfaction question at the month 12 visit. Safety Assessment: Safety assessment include: Treatment emergent adverse events (TEAEs) Focused physical examination (PE) Safety Objectives and The safety objective of the study is to evaluate the safety of abobotulinumtoxinA in **Endpoints:** the treatment of glabellar lines. The safety endpoint will include the incidence and severity of treatment emergent adverse events (TEAEs) throughout the study. Other Assessments: Other assessments include: **Pregnancy Test** Principal statistical method: The primary objective of the study will be evaluated by calculating the proportion of subjects that respond "Highly satisfied" or "Satisfied"



| SYNOPSIS | |
|---|---|
| Clinical Study Title: Dysport Efficacy and Measured Satisfaction (DREAM) Study: A Multicenter, Open-Label, Interventional Study to Evaluate Subject Satisfaction of AbobotulinumtoxinA Treatments in Moderate to Severe Glabellar Lines | |
| | The aim is to show that the confidence interval is above 50%, i.e. the majority of subjects are satisfied. |
| | Incidence and severity of TEAEs will be presented descriptively. |







GALDERMA 43USD480256linical Standar Protocycl Describ DBFA MREAM study

Doc id

**MA-38095** 



GALDERMA 43USD480256linical Standar Protocycl Describ DBFA Drendem study

**MA-38095** 

Doc id





## LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Term |
|---|---|
| °C | Degrees Celsius |
| AbobotulinumtoxinA | Commercially available DYSPORT® |
| AE | Adverse Event |
| approx | Approximately (or use 'about', not C. or ca.) |
| CDMS | Clinical Data Management |
| CPM | Clinical Project Manager |
| CRA | Clinical Research Associate |
| CRF/eCRF | Case Report Forms/electronic Case Report Forms |
| CRO | Contract Research Organization |
| DC | Discontinuation |
| DMP | Data Management Plan |
| e.g. | For Example (Latin: exempli gratia) |
| ET | Early Termination |
| etc | Et cetera |
| FDA | Food and Drug Administration |
| FSFV | First Subject First Visit (date of first subject included i.e., informed consent signature) |
| GL | Glabellar line |
| GCP | Good Clinical Practice |
| HIPAA | Health Insurance Portability and Accountability Act of 1996 |
| ICH | International Conference on Harmonisation |
| ID | Identity |
| i.e. | That is (Latin: id est) |
| IRB | Institutional Review Board |
| ITT | Intent-to-treat |
| IUD | Intrauterine Device |
| LOCF | Last Observation Carried Forward |
| LSFV | Last Subject First Visit (date of last subject included i.e., informed consent signature) |
| LSLV | Last Subject Last Visit (date of last subject's last study visit) |
| MD | Medical Doctor |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mL | Milliliter |
| N/A | Not Applicable |
| OTC | Over-the-Counter |



| Abbreviation | Term |
|--------------|-----------------------------------------------|
| p | Page(s) |
| PE | Physical Examination |
| PP | Per-Protocol |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| TOC | Table of Contents |
| TEAE | Treatment-emergent Adverse Event |
| UPT | Urine Pregnancy Test |
| US | United States |
| USP | United States Pharmacopeia |



#### 1 BACKGROUND AND RATIONALE

| 1.1 Medical Background and Short Rationale for the Clinical Study |
|---|
| Botulinum toxin (BoNT) is a potent neurotoxic protein produced by the Gram-positive anaerobic bacterium, Clostridium botulinum. The molecule is produced naturally by these bacteria together with a series of accessory proteins, forming what is termed the "toxin complex". The neurotoxin is the cause of the severe and potentially fatal disease of botulism. In addition, the protein is used in very small quantities as a treatment modality for aesthetic and medical indications, many of which are characterized by increased muscle activity. |
| In the early 1990s, patients treated with BoNT-A for blepharospasm were observed to lose their frown lines, <sup>1, 2</sup> and since publishing these observations, the use of BoNT-A in the aesthetic setting has accelerated. Injectable BoNT-A products have been investigated for multiple aesthetic indications in attempts to reverse the appearance of aging, especially in the facial region. <sup>1</sup> |

AbobotulinumtoxinA (Dysport) was approved by the United States Food and Drug Administration (FDA) in 2009. AbobotulinumtoxinA is indicated for the temporary improvement in the appearance of moderate to severe GL associated with procerus and corrugator muscle activity in adult patients less than 65 years of age.

The rationale for the current study is to evaluate subject satisfaction, efficacy, and safety of of abobotulinumtoxinA administered in the glabellar region. The aim is for the Sponsor to better understand the subject's needs and expectations with respect to abobotulinumtoxinA treatment and the treatment regimen.

#### 1.2 Drug Profile

AbobotuliniutoxinA contains a neurotoxin complex that is produced by fermentation of Clostridium botulinum bacteria toxin type A, Hall strain. This haemagglutinin complex is





#### 2 CLINICAL STUDY OBJECTIVES AND CLINICAL HYPOTHESIS

## 2.1 Clinical Study Objectives

The objectives of this study are to evaluate subject satisfaction, efficacy, and safety after abobotulinumtoxinA treatment every six months (twice yearly).



#### 2.1.1 Primary Efficacy Objectives and Endpoints

The primary objective of the study is to evaluate subject satisfaction after abobotulinumtoxinA treatment every six months (twice yearly).



The primary endpoint will evaluate the proportion of subjects satisfied ("highly satisfied" or "satisfied") with the treatment results assessed by the satisfaction question at the month 12 visit.





#### 2.1.3 Safety Objectives and Endpoints

The safety objective of the study is to evaluate the safety of abobotulinumtoxinA in the treatment of glabellar lines.

The safety endpoint will include the incidence and severity of treatment emergent adverse events (TEAEs) throughout the study.

## 2.2 Clinical Hypothesis

The clinical hypothesis of the study is that a majority of subjects will be highly satisfied or satisfied with the treatment results using abobotulinumtoxinA every 6 months.

#### 3 OVERALL CLINICAL STUDY DESCRIPTION

This is a multicenter, open-label, interventional, phase 4 study to assess subject satisfaction with a twice-yearly abobotulinumtoxinA treatment regimen.

| Following signature of informed consent and the screening process, eligible subjects will be treated |
|---|
| at the baseline visit (Day 0) with abobotulinumtoxinA in the glabellar region. Subject |
| will be re-treated at the month 6 visit, |
| Subjects will be monitored for up to 13 months following the initial treatment at baseline |



#### 4 CLINICAL STUDY DURATION AND TERMINATION

The planned clinical study duration (from FSFV to LSLV) is approximately 15 months. The date of end of the clinical study is defined as the date of the last visit of the last subject.



#### 5 SELECTION AND DISPOSITION OF CLINICAL STUDY POPULATION

5.1

## 5.2 Clinical Study Population Characteristics

In order to be eligible for the clinical study, subjects must fulfill all of the following criteria. These criteria are applicable at screening/baseline unless specified.

#### 5.2.1 Inclusion Criteria

1. Male or female, 18 to 65 years of age.



4. Female of non-childbearing potential (i.e., post-menopausal [absence of menstrual bleeding for 1 year prior to screening, without any other medical reason], or has undergone hysterectomy or bilateral oophorectomy).

or

Female of childbearing potential with a negative urine pregnancy test at screening/ baseline, and agrees to use an acceptable, reliable and approved contraceptive method for the duration of enrollment in the study. Male subjects do not require birth control measures.





## **5.2.2** Exclusion Criteria

- 1. Botulinum toxin treatment in the face within 9 months prior to the screening/baseline visit.
- 2. Known allergy or sensitivity to any component of the study product, or allergy to cow's milk protein.







12. Receipt of any investigational drug or device within 30 days prior to study treatment, from a previous clinical study.



#### 5.3 Medical History

Relevant history of surgical events and medical conditions shall be documented in the electronic case report form (eCRF) using medical terminology.

#### 5.4 Previous and Concomitant Therapies

#### **5.4.1** Definition

Previous therapies are defined as therapies that have been stopped within the 4 weeks preceding the screening visit or within timeframes specified in the inclusion/exclusion criteria.

Concomitant therapies are defined as follows:

- any existing therapies ongoing at the time of the screening visit,
- any changes to existing therapies (such as changes in dose or formulation) during the course of the clinical study, or
- any new therapies received by the subject since the screening visit.








#### 5.5 Procedures/Reasons for Subject Discontinuation

An Investigator may decide to discontinue a subject from the clinical study for safety reasons.

Although the importance of completing the entire clinical study should be explained to the subject by the clinical study personnel, any subject is free to discontinue participation in this clinical study at any time and for whatever reason, specified or unspecified, and without any prejudice. No constraints are to be imposed on the subject, and when appropriate, a subject may be treated with other conventional therapy when clinically indicated.



All discontinuations and the reason for discontinuation are to be documented by the Investigator on the exit form. For discontinuation due to an AE, the AE form is to be completed. The Investigator should also ensure that the subject receives suitable therapy for the AE.



Pregnancies occurring during the screening period are considered screen failures; they should be recorded as such in the eCRF and no pregnancy form is to be completed. In case of a pregnancy occurring after the baseline visit, follow the procedures described in Section 8.2.1.2.3. The subject





may remain in the study, but no invasive procedure should be conducted (e.g. no sample taken for lab test).

The Sponsor may also decide to prematurely terminate or suspend a subject's participation in the clinical study.



#### 6 CLINICAL SUPPLIES

Details of the drug composition and excipients are provided in the current US prescribing information.<sup>3</sup>



#### 6.1.2 Subject Identification Number (SIN)

Each study participant who has signed the ICF will be entered into the eCRF system and a subject number will be assigned via the eCRF system.



All subjects who have signed the ICF should be listed. Sufficient information to link the eCRF to the medical records should be recorded in the source documentation.

For the duration of the entire study, the subject will be identified using the subject number for all documentation and discussion.

## 6.1.3 Method of Treatment Assignment

Not applicable; this is an open-label study.

#### **6.1.4** Kit Number/Randomization Number

Not applicable; this is an open-label study.

| 6.1.5 |
|-------|







## 6.2 Study Drug(s) Packaging and Labeling

The carton will contain a label indicating the protocol number and that the product is for a clinical study.

#### 6.3 Supplies Management

#### 6.3.1 Accountability

Upon receipt of the study drug(s), the Investigator or designee will maintain accurate records of the study drug(s) delivery to the clinical study center, the inventory at the clinical study center, the use by each subject, the reconciliation of all study drug(s) received from the Sponsor's designee, and the return to the Sponsor's designee for disposal of used and unused study drug(s).

All study drug(s) sent to the Investigator/Institution will be accounted for and no unauthorized use is permitted.

#### 6.3.2 Storage of Study Drug(s)

Study drug(s) must be stored in a safe and secure area with restricted access, under the storage conditions specified by the Sponsor (see Table 3).



#### 6.3.3 Dispensing and Return

All study drug must be inventoried and a record of the dispensing for each subject must be appropriately documented by the Investigator or designee. Any dispensing errors must be reported to the Sponsor/CRO and properly documented.

In the event of early termination/suspension of the clinical study, a rapid recall of study drug(s) will be initiated.

#### 6.3.4 Treatment Compliance Management and Record

The treatment is an injection administered by the Investigator. It will be recorded in the eCRF that the injection has been administered. No other measurements of treatment compliance will be made.



#### **6.4** Dose Modification

Dose modifications are not permitted.

#### 6.5 Blinding

Not applicable; this is an open-label study.



## 7 EFFICACY ASSESSMENTS

7.1 Overall Subject Satisfaction by Direct Questioning









#### 8 SAFETY ASSESSMENTS

A safety assessment will be conducted for all subjects at the screening visit (from the Informed consent signature) and at subsequent visits as outlined in the schedule of assessments (Table 2). Safety parameters include an evaluation of AES and focused physical examination findings.

#### 8.1 Focused Physical Examination

At all study visits (prior to treatment, as applicable), the Investigator or designee will perform a physical examination of the subject that includes the face, head, and neck. Further details are provided in Appendix 4.



The Investigator may choose to investigate any other sign that he/she observes during the physical examination and should assess all abnormal findings for clinical significance.

Clinically significant abnormal findings at the screening/baseline visit are exclusionary, and the subject should not be enrolled in the study. If the abnormality is not clinically significant, capture it as medical history.

For any clinically significant changes from the screening/baseline visit, an AE is to be recorded.

#### 8.2 Adverse Events

AEs are to be monitored throughout the course of the clinical study from the time the informed consent form has been signed. All AEs are to be reported on the AE form of the eCRF with complete information as required.

If AEs occur, the main concern shall be the safety of the subjects. At the time of the ICF signature, each subject must be provided with the name and phone number of clinical study center personnel for reporting AEs and medical emergencies.

#### 8.2.1.1 Definitions

#### 8.2.1.1.1 Adverse Events (AE)

According to ICH E2A, an AE is any untoward medical occurrence in a patient or a clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended


sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (study) product, whether or not related to the medicinal (study) product.

Thus any new sign, symptom or disease, or any clinically significant worsening of an existing sign, symptom or disease (including new episodes of a chronic disease [e.g., hay fever, allergy]) compared to the condition at the first visit, should be considered as an AE. Lack of efficacy is not considered as an AE.

### Notes:

- There should be an attempt to report a diagnosis rather than the signs, symptoms or abnormal laboratory values associated with the report of an AE. However, a diagnosis should be reported only if, in the Investigator's judgment, it is relatively certain. Otherwise, symptoms, signs, or laboratory values should be used to describe the AE.
- Pregnancy is not to be considered as an AE; however, is an important medical event that must be monitored as described in Section 8.2.1.2.3.

### 8.2.1.1.2 Treatment Emergent Adverse Events (TEAE)

A TEAE is an event that emerges during treatment, having been absent pre-treatment, or worsens relative to the pretreatment state.

Investigators are responsible for monitoring, recording, and reporting all AEs that occur during the study as described. TEAEs will be delineated from AEs following database lock.

# 8.2.1.1.3 Serious Adverse Events (SAE)

An SAE is any untoward medical occurrence that at any dose:

- Results in death,
- Is life-threatening,
- Requires inpatient hospitalization or prolongation of existing hospitalization,
- Results in persistent or significant disability/incapacity, or
- Is a congenital anomaly/birth defect.

Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, they may jeopardize the safety of the subject, and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasia, or convulsions that do not result in hospitalization.

Note: The term "life-threatening" refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe.



Inpatient hospitalization is considered to have occurred if the subject has had to stay for a night at the hospital. The criterion for prolongation of hospitalization is also defined as an extra night at the hospital. Hospitalization may not constitute sufficient grounds to be considered as an SAE if it is solely for the purpose of a diagnostic test(s) (even if related to an AE), elective hospitalization for an intervention that was already planned before subject enrolment in the clinical study, admission to a day-care facility, social admission (e.g., if the subject has no place to sleep), or administrative admission (e.g., for a yearly examination).

### 8.2.1.1.4 Unexpected Adverse Drug Reaction

An unexpected adverse drug reaction is defined as an adverse reaction, the nature or severity of which is not consistent with the applicable study product information (e.g., medicinal package insert/summary of product characteristics for an approved study product).

# 8.2.1.1.5 Adverse Event Reporting Period

The clinical study period during which AEs must be reported is the period from when the subject signed the ICF to the end of the subject's participation.

The Sponsor should be informed if the Investigator becomes aware of any unusual safety information or any safety information that appears to be drug-related involving a subject who has participated in a clinical study, even after a subject has completed the clinical study.

### 8.2.1.1.6 *Severity*

Severity is a clinical determination of the intensity of an AE and not the severity of a disease.

The Investigator is to classify the intensity of AEs using the following definitions as a guideline. For this classification, the Investigator will take into account the possible range of the intensity of the event and report the grade of intensity which is the most appropriate according to his/her medical judgment.

**Mild** Awareness of signs or symptom, but easily tolerated.

Moderate Discomfort, enough to cause interference with usual activity.

Severe Incapacitating with inability to work or perform usual activity.

# 8.2.1.1.7 Relationship to the Study Product and/or Clinical Study Procedure

The Investigator is to determine whether there is a reasonable causal relationship between the occurrence of the AE and exposure to the study product and/or clinical study procedure.

Medical judgment should be used to determine the relationship, considering all relevant factors including the pattern of reaction, temporal relationships, relevant medical history, and confounding factors such as co-medication or concurrent diseases.



The expression "reasonable causal relationship" is meant to convey in general that there are facts or arguments to suggest a causal relationship (ICH E2A, Section IIIA 1).

The relationship assessment for an AE is to be completed using the following definitions as a guideline:

### **Reasonable Possibility:**

According to the reporting Investigator, there is a reasonable possibility (i.e., suggestive evidence or arguments) that there is a causal relationship irrespective of the dose administered between:

- The study product and the AE.
- The clinical study protocol procedure (injection related trauma, etc.) and the AE.

A two-point scale (Yes or No response) shall be used for the causality assessment. The Investigator shall be asked to indicate a response to each of the following questions in the eCRF:

- "Do you consider that there is a reasonable possibility that the event may have been caused by the study product?", and
- "Do you consider that there is a reasonable possibility that the event may have been caused by the study product injection procedure?"

If any of these questions is answered Yes, the AE is considered related.

## No Reasonable Possibility:

No suggestive evidence or arguments can be identified regarding a causal relationship between the study product or the clinical study protocol procedure and the AE.

### 8.2.1.2 Reporting Procedures

### 8.2.1.2.1 Procedures for Reporting Adverse Events

The collection of AEs is from the time that a subject signs the ICF to their final visit.

At each post-enrollment visit, the Investigator (or sub-Investigator) will question the subject about AEs using an open non-persuasive question to elicit reporting of AEs, for example "Have you noticed any change in your health since the last visit?" Directed questioning and examination will then be performed as appropriate.

Any AE occurring during the AE reporting period, whether it is related to the study product or not, will be recorded immediately in the source document, and described on the AE form of the eCRF along with the date of onset, severity, relationship to the study product, and outcome, without omitting any requested and known information. Additional information will be requested under certain circumstances.



Adverse Events (AEs) assessed as related to the treatment or study procedure will be monitored until they have resolved or reached a stable condition. Other AEs will be monitored until the last visit if they have not resolved or reached a stable condition.

The Investigator will obtain and maintain in the subject's files all pertinent medical records, information and medical judgment from colleagues who assisted in the treatment and follow-up of the subject. If necessary, the Investigator will contact the subject's personal physician or hospital staff to obtain further details.

For SAEs (see Section 8.2.1.2.2) and pregnancies (see Section 8.2.1.2.3), the Sponsor is to be informed immediately by e-mail. The event must be reported by e-mail to the Safety Mailbox within 24 hours of receipt of the information (contact details in Section 8.2.1.2.2).

# 8.2.1.2.2 Procedure for Reporting a Serious Adverse Event

For a SAE occurring during the period of the clinical study, regardless of whether it is related to the treatment or not, and of whether it is expected or not, the Investigator must do the following:

- 1. Take prompt and appropriate medical action, if necessary. The safety of the subject is the first priority.
- 2. Ensure that the event is classified as an SAE (Section 8.2.1.1.3).
- 3. Complete the AE form provided in the eCRF as fully as possible.

Print and complete the SAE form. E-mail the completed form, accompanied by any other relevant information or anonymized medical records (e.g., laboratory test results) within 24 hours of receipt of the information to the Safety Mailbox listed below. The demographics, medical history, drugs/therapies form, medical and surgical procedures form, and AE pages of the eCRF must be completed and available for review in the EDC system at the time of the report.

- 4. Immediately send the completed SAE report form to the Safety Mailbox via e-mail and discuss further actions to be taken.
- 5. Monitor and record the progress of the event until it resolves or reaches a clinically stable outcome, with or without sequelae. For all additional follow-up evaluations, send by e-mail all additional follow-up information on the SAE to the Safety Mailbox within 24 hours of receipt of the updated information. SAEs will be monitored until the Investigator and Sponsor agree that the event is satisfactorily resolved.
- 6. Obtain and maintain in his/her files all pertinent medical records, information, and medical judgments from colleagues who assisted in the treatment and follow-up of the subject. If necessary, contact the subject's personal physician or hospital staff to obtain further details.



- 7. Inform the Sponsor of the final outcome of the event. Send a revised or updated SAE form and AE form, if appropriate to the Safety Mailbox.
- 8. Prompt notification of SAEs by the Investigator to the Sponsor is essential so that legal obligations and ethical responsibilities towards the safety of subjects are met. The Sponsor has a legal responsibility to notify both the local regulatory authority and other regulatory agencies about the safety of a product under clinical investigation. The Sponsor will comply with country specific regulatory requirements relating to safety reporting to regulatory authorities, Institutional Review Boards (IRBs), and Investigators. Investigator safety reports are prepared for Suspected Unexpected Serious Adverse Reactions (SUSARs) according to local regulatory requirements and the Sponsor policy and are forwarded to Investigators as necessary. An Investigator who receives an Investigator safety report describing a SAE(s) or other specific safety information (e.g., summary or listing of SAEs) from the Sponsor will file it with the prescribing information and will notify the IRB, if appropriate according to local requirements.
- 9. Comply with the applicable regulatory requirement(s) related to the reporting of SAEs to the IRB.

## 8.2.1.2.3 Procedures for Reporting Pregnancies

Any pregnancy occurring during the clinical study, where the fetus could have been exposed to the study product, must be monitored until its outcome in order to ensure the complete collection of safety data.

Pregnancies occurring during the screening period are considered as screening failures; they are recorded as such in the eCRF and no pregnancy form is to be completed.

If a subject becomes pregnant after the screening period, the Investigator is to do the following:

- 1. The subject does not need to be withdrawn from the clinical study, i.e. she may continue to attend the planned study visits, but no invasive procedure should be conducted (e.g. no sample taken for lab test).
- 2. Complete the Pregnancy Surveillance form Part I: History and Start of Pregnancy, as fully as possible. Send by e-mail this pregnancy form along with the exit form (if applicable) within 24 hours of receipt of the information to the Safety Mailbox listed above (see Section 8.2.1.2.2).
- 3. Monitor and record the progress of the pregnancy until its outcome. Contact the subject's regular physician (general practitioner or gynecologist) or hospital staff to obtain further details and ask regular follow-up information.
- 4. Inform the Sponsor of the progress by tri-monthly updates until the final outcome of the pregnancy by completing the Pregnancy Surveillance form Part I. For all the additional evaluations, send by e-mail the additional follow-up information to the Safety Mailbox within 24 hours of receipt of the information. If the subject can no longer be reached (lost to



follow-up), documentation of the non-response/contact with two phone calls and a letter (certified with return receipt) is required.

- 5. At the outcome of the pregnancy, complete the Pregnancy Surveillance form Part II: Course and Outcome of Pregnancy, as fully as possible. Inform the Sponsor by sending this pregnancy form to the Safety Mailbox within 24 hours of receipt of the information.
- 6. If the pregnancy leads to an abortion (voluntary abortion, spontaneous abortion or therapeutic abortion), *in utero* death or congenital anomaly, follow the procedure for declaration of an SAE (see Section 8.2.1.2.2).



For all women of childbearing potential a urine pregnancy test will be performed prior to treatment at screening/baseline and month 6, and month 12 (if optional re-treatment is performed). A negative pregnancy test is required for study inclusion. The result will be documented.

### 8.4 Appropriateness of Measurements

The subject satisfaction question and questionnaire are tools that have been developed in order for the Sponsor to better understand the subject's needs and expectations with respect to abobotulinumtoxinA treatment and the treatment regimen.





### 9 CLINICAL STUDY VISITS DESCRIPTIONS AND PROCEDURES

# 9.1 Description of Clinical Study Visits

Please refer to the schedule of assessment table (Table 2).

A written, signed ICF (inclusive of HIPAA and photo consent) must be obtained prior to performing any clinical study-related evaluations and/or procedures. The subject must be provided with a fully completed, dated and signed copy.




















## 10 STATISTICAL METHODS PLANNED



10.1.2.4 Safety Population

The safety population includes all subjects who were administered the study product.



### 10.1.2.5 Imputation of Missing Data

All analyses will be carried out based on the observed cases (OC). However, if there are a substantial amount of missing data for the primary efficacy endpoint, a sensitivity analysis to assess the impact of the missing data might be done by using, for example, the hot deck method.

# 10.1.3 Data Presentation and Graphics

Subject disposition, completion and discontinuation by study visit, protocol deviations, demographics and baseline characteristics, medical history, medical and surgical procedures, prior and concomitant medications, will be summarized.



### 10.1.3.1 Safety

A summary of all AEs will be provided, which will include:

- number of subjects who did not have an AE
- number of subjects with at least one AE and number of events
- number of subjects with at least one TEAE and number of events
- number of subjects with at least one related TEAE and number of events
- number of subjects with at least one TEAE by causality
- number of subjects with at least one TEAE by maximum intensity
- number of subjects with at least one TEAE leading to discontinuation
- number of subjects with at least one serious TEAE.

All TEAEs, treatment emergent SAEs, TEAEs by maximum intensity, TEAEs by causality, TEAEs by maximum intensity and causality, and TEAEs leading to discontinuation will be summarized



by SOC and PT including number of subjects with at least one event, percentages, and number of events. All related TEAEs will also be summarized by time to onset and duration.

The results of the urine pregnancy tests will be listed.

### 10.1.4 Withdrawals and Deviations

All withdrawn subjects will be listed individually, including at least subject number, date and reason for withdrawal, and last visit performed.







10.3

# 11 TRAINING / MONITORING / DATA MANAGEMENT / QUALITY ASSURANCE

### 11.1 Personnel Training

Investigators and other responsible persons should be listed together with their function on the delegation log. Study staff shall provide a curriculum vitae or equivalent, as appropriate.

It is the responsibility of the PI to ensure that all personnel involved in the study are fully informed of all relevant aspects of the study, including detailed knowledge of and documented training in all procedures to be followed.

### 11.2 Clinical Monitoring

The conduct of the clinical study will be closely monitored by representatives of the Sponsor to verify adherence to the clinical study protocol, ICH-GCP guidelines, and applicable SOPs.

The Investigator will allow the CRO/Sponsor's representatives, to have direct access to all clinical study records, CRFs, corresponding subject medical records, study product(s) dispensing records, and any other documents considered source documentation. Additionally, the CRO/Sponsor representative is to have access to the study product storage area and clinical study facilities.

The Investigator also agrees to assist the representative if required.

### 11.3 Data Management

All data management procedures will be detailed in a Data Management Plan (DMP).

# 11.4 Quality Assurance / Audit / Inspection

The clinical study is conducted under the sponsorship of the Sponsor in compliance with the applicable international and local regulatory requirements as well as applicable ICH guidelines and in accordance with the SOPs for clinical study conduct and monitoring from the Sponsor and/or the Contract Research Organization (CRO).

Audits of clinical study centers may be conducted by the Sponsor/CRO representatives, and inspection may be performed by Regulatory Authority inspectorates or IRBs/IECs before, during, or after the clinical study.





The Investigator will allow and assist the CRO/Sponsor's representatives, IRBs/IECs and any regulatory agency to have direct access to all requested clinical study-related records.

For the audits performed by, or on behalf of, the Sponsor auditors, audit certificate(s) will be provided by Quality Assurance.





### 12 ETHICS AND GENERAL CLINICAL TRIAL CONDUCT CONSIDERATIONS

### 12.1 Institutional Review Board (IRB)

This clinical study protocol and all amendments will be reviewed and approved by the appropriate IRBs.

### 12.2 Ethical Conduct of the Clinical Study

This clinical study will be conducted in accordance with the protocol, the HELSINKI declaration (1964) and subsequent amendments, and the ICH GCP, and in compliance with applicable regulatory requirements.

### 12.3 Subject Information and Consent

All subjects who participate in this clinical study are required to be fully informed about the clinical study in accordance with GCPs guidelines, federal regulations, HIPAA, and guidelines and in accordance with local requirements.

The ICF (inclusive of HIPPA and photo consent), approved by an IRB/IEC, will be fully explained to the subject. The subject must agree to photo consent in order to participate in the clinical study.

Prior to enrollment into the clinical study, the subject and the PI or designee must sign and date the consent form(s). The Investigator is responsible for maintaining each subject's consent form(s) in the Investigator's site file and providing each subject with a copy of the signed and dated consent form(s).

### 12.4 Protection of Personal Data

The completion of the study involves the gathering and processing of Personal Data as specified in the Regulation (EU) 2016/679 on the protection of individuals with regard to the processing of personal data and on the free movement of such data. For the purposes of the study, Sponsor will be considered the Data Controller, and Principal Investigator and Institution will both be considered Data Processors.

All processing of Personal Data must be carried out in accordance with national legislation concerning the protection of Personal Data. The Institution and Principal Investigator are responsible for complying with all requirements pursuant to national legislation in the country in which the Institution and Principal Investigator are located.

The Sponsor shall, to the extent feasible, protect study subject identifier information.

The Institution and Principal Investigator are jointly responsible for obtaining the appropriate informed consent of each subject for the processing of Personal Data required in order to complete



the study. Such consent shall include the consent to the transfer of Personal Data to government authorities located in countries outside the US.

The Institution and Principal Investigator are jointly responsible for providing sufficient information to all subjects to enable them to give their informed consent not only to the participation in the study, but also to the processing of Personal Data. Such information includes information regarding the purposes of the processing, the length of time during which Personal Data will be stored, the right of access to stored Personal Data and the right to correction or purging of incorrect or obsolete Personal Data. A subject may also withdraw his or her consent at any time. A subject who withdraws his or her consent to the processing of Personal Data must be considered to have withdrawn from the study but the data collected until the consent was withdrawn may be used in the statistical analyses.

All collection, processing and analyses of protected health information, personal data or similar will be conducted in compliance with applicable local, national and international rules, regulations and guidelines.

### 12.5 Contractual Requirements

A contractual agreement will be signed between the CRO/Sponsor and each Investigator/Institution. This document will contain supplementary information, including financial terms, confidentiality, the clinical study schedule, third party responsibility, and publication rights.

### 12.6 Data Collection and Archiving

### 12.6.1 Data Collection

The Investigator must maintain all required records for all subjects. Data for this clinical study will be recorded in the subject's source documents and in the eCRFs provided by the Sponsor. All data should be recorded in the eCRFs completely and promptly.

### 12.6.2 Source Documentation

The Investigator must keep accurate separate records (other than the eCRFs) of all subject visits, being sure to include all pertinent clinical study-related information. A statement should be made indicating that the subjects have been included in this clinical study and have provided signed written Informed Consent. All AEs must be thoroughly documented.

Results of any diagnostic tests conducted during the clinical study should also be included in the source documentation.



### 12.6.3 Archives

All pertinent data, samples, photographs, correspondence, and reports, the original or amended clinical study protocol, and all other material relating to the clinical study will be maintained securely in Sponsor/CRO/Investigator/Institution archives for the legally required duration for archiving.

The Investigator/Institution should maintain the essential clinical study documents as specified in Section 8 of ICH-GCP, and according to the applicable regulatory requirements.

The Investigator/Institution should take measures to prevent accidental or premature destruction of these documents.

If the Principal Investigator retires, relocates, or withdraws from the responsibility of keeping the clinical study records for any other reasons, custody must be transferred to a person who will accept the responsibility. The Sponsor/CRO must be notified in writing of the name and address of the new custodian.

### 12.7 Insurance

A certificate attesting Third Party coverage of CRO/Sponsor will be provided upon request.



<sup>&</sup>lt;sup>a</sup> Defining the role of authors and contributors, compiled by the International Committee of Medical Journal Editors (ICMJE) (http://www.icmje.org).







### 13 LITERATURE REFERENCE LIST

- 1. Monheit GD, Pickett A. AbobotulinumtoxinA: A 25-Year History. Aesthet Surg J. 2017 May 1;37(suppl 1):S4-S1.
- 2. Carruthers J, Carruthers A. The evolution of botulinum neurotoxin type A for cosmetic applications. J Cosmet Laser Ther. 2007 Sep;9(3):186-92.
- 3. Rzany B, Dill-Müller D, Grablowitz D, et al. Repeated botulinum toxin A injections for the treatment of lines in the upper face: a retrospective study of 4,103 treatments in 945 patients. Dermatol Surg. 2007 Jan;33(1 Spec No.):S18-25.
- 4. DYSPORT® (abobotulinumtoxinA) for injection, for intramuscular use [Prescribing Information]. Wrexham, UK: Ipsen Biopharm Ltd: 12/2016.

| 5. |
|----|


































# SIGNATURES PAGE

